CLINICAL TRIAL: NCT05405049
Title: Intraperitoneal Instillation and Wound Infiltration Compared With Intrathecal Morphine for Postcesarean Section Analgesia : A Prospective Randomized Controlled Double- Blind Trial
Brief Title: Compared With Different Method for Postcesarean Section Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Aysenur Dostbil, Clinical Professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B.30.2.ATA.0.01.00/339
Record Dates: First submitted 2022-05-24; First posted 2022-06-03 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2022-06

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Bupivacaine; Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group intraperitoneal instillation of local anesthetic + local anesthetic infiltration (IPLA+ LWI) (Active Comparator): local anesthetic infiltration into all layers of the anterior abdominal wall and peritoneal instillation
  Interventions: Drug: Bupivacain
- Group morphine ( M ) (Active Comparator): intrathecal injection of morphine with local anesthesic
  Interventions: Drug: Morphine hydrochloride

INTERVENTIONS:
Drug: Morphine hydrochloride — Group M will be given a 0.5% Bupivacain Dosage Regimen with weight and height adjustment+15 μg fentanyl +150 μg morphine intrathecally.
  Other Names: Bupivacaine; fentanyl
  Arms: Group morphine ( M )
Drug: Bupivacain — Group LWI+IPLA will given 30 ml %0,5 bupivacaine+%2 lidocaine infiltration and instillation
  Other Names: lidocain; fentanyl
  Arms: Group intraperitoneal instillation of local anesthetic + local anesthetic infiltration (IPLA+ LWI)

SUMMARY:
The aim of this study is compare the efficacy of local anesthetic infiltration into all layers of the anterior abdominal wall and peritoneal instillation and intrathecal injection of morphine with local anesthesic to reduce pain in women undergoing elective cesarean section under spinal anesthesia. The primary outcome is to compare the total amount of opioids consumed in the first 24 hours postoperatively.

Secondary purpose; Pain scores at 2,4,6,12,and 24 hours during movement ( moving back and forth in bed ) and rest ( lying motionless in bed )

DETAILED DESCRIPTION:
This prospective randomized double-blind study will be planned on 46 pregnant women aged 18-50 who will undergo cesarean section with Pfannenstiel incision under spinal anesthesia with American Society of Anesthesiologists Classification (ASA) II,fullterm singular pregnancy after receiving the approval of the ethics committee of Ataturk University Medical Faculty Hospital and written approval of the patients

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* 18-50 age
* ASA II
* Fullterm singular pregnancy

Exclusion Criteria:

* Neuraxial anesthesia is contraindicated,
* Allergy to the drugs to be used in the study,
* Refused to participate in the study,
* BMI>35 kg/m2
* ASA≥3
* Diabetes
* Preeclampsia,
* Cardiovascular disease
* Chronic pain and neuropathic pain,
* Given opioids in the operation due to intraoperative pain,
* Switched to general anesthesia,
* Excessive bleeding during the operation,
* Uterine atony
* Drain placed in the area to be infiltrated,
* History of drug addiction and psychiatric illness,
* Understand Visual analog pain scale

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2022-06-16 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2023-11-11 (Actual)

PRIMARY OUTCOMES:
The primary outcome is to compare the total amount of opioids consumed in the first 24 hours postoperatively. | postoperative 24 hours
  The primary outcome is to compare the total amount of opioids consumed in the first 24 hours postoperatively.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) (0-10) at 2,4,6,12 and 24 hours postoperatively | 2,4,6,12,and 24 hours postoperatively
  The VAS is a validated.Possible scores range from 0 (no pain) to 10 (worst possible pain)

CONTACTS AND LOCATIONS:
Overall Officials: ayşenur dostbil, prof, Principal Investigator — Department of Anesthesiology and Reanimation.Ataturk Universty School of Medicine
Locations (1):
- Atatürk üniversty medicine school, Erzurum, YAKUTİYE, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No